CLINICAL TRIAL: NCT02678650
Title: Department of Anesthesiology, Beijing Anzhen Hospital, Capital Medical University
Brief Title: MicroRNA Mediates Volatile Anesthetics Preconditioning Induced Artery Protection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liang Zhang (Other)
Responsible Party: Sponsor-Investigator, Liang Zhang, Principal Investigator, Beijing Anzhen Hospital
Organization: Beijing Anzhen Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015017X
Record Dates: First submitted 2016-01-23; First posted 2016-02-10 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Coronary Artery Bypass Graft Triple Vessel
Keywords: Volatile Anesthetics; MicroRNA; Off-pump Coronary Artery Bypass Surgery; Internal Mammary Artery; Ascending Aorta

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- volatile anesthetics group (Experimental): 10min after intubation, begin to sevoflurane wash-in / wash-out operation: sevoflurane administration was interrupted for at least 10 min, by washout with a high fresh gas flow (10 l/min) to achieve a MAC value below 0.2. Following the interruption, sevoflurane was again washed in with a high fresh gas flow (6 l/min) to achieve 1 MAC end-tidal concentration as soon as possible, and repeated twice periods of 10 minutes. Discontinuation of the halogenated agent for at 15 minutes during the last wash out time.
  Interventions: Drug: volatile anesthetics(isoflurane)
- propofol intravenous anesthesia group (Placebo Comparator): propofol infusion 3-5μg / kg / h
  Interventions: Drug: propofol intravenous anesthesia

INTERVENTIONS:
Drug: volatile anesthetics(isoflurane) — volatile anesthetics wash-in / wash-out operation
  Arms: volatile anesthetics group
Drug: propofol intravenous anesthesia — propofol infusion 3-5μg / kg / h
  Arms: propofol intravenous anesthesia group

SUMMARY:
It has been reported that volatile anesthetics preconditioning mediates protection of organ via microRNA. We want to study on the effects of isoflurane preconditioning on expression of microRNA and mRNA in the specimens of internal mammary artery and ascending aorta.

DETAILED DESCRIPTION:
1. Sixty patients scheduled for off-pump coronary artery bypass surgery were randomly assigned to isoflurane wash-in/wash-out group(S-I group, n=30)or propofol intravenous anesthesia group(P group, n=30).
2. Anesthesia and monitoring method All patients were monitored according to the American Society of Anesthesia guidelines and received standard general induction of anesthesia.
3. SI group:10min after intubation,begin to isoflurane wash-in/wash-out operation:isoflurane administration was interrupted for at least 10 min,by washout with a high fresh gas flow(10 l/min)to achieve a MAC value below 0.2. Following the interruption,sevoflurane was again washed in with a high fresh gas flow(6 l/min)to achieve 1 MAC end-tidal concentration as soon as possible,and repeated twice periods of 10 minutes.Discontinuation of the halogenated agent for at least 15 minutes during the last wash out time.
4. P Group:propofol infusion 3-5μg/kg/h.
5. When isoflurane inhaled anesthetic,propofol are stopped infusion.If during this interruption the BIS value increased to>50,0.5 mg/kg propofol was administered repeatedly in boluses until the BIS value have returned to<50.

6.1h after isoflurane preconditioning,specimens of internal mammary artery(surplus arterial tissue is obtained from the repair internal mammary artery)and ascending aorta(the stump after ascending aortic punch)will be saved, and before isoflurane preconditioning,1h,3h,5h after isoflurane preconditioning, central venous blood samples will also be drawn.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* written informed consent;
* scheduled procedures;
* planned isolated OPCABG(multiple bypass are allowed; planned combined intervention such as CABG plus valve surgery are not allowed);
* ejection fraction> 50%;
* NYHA class Ⅱ~Ⅲ;
* serum creatinine <150μmol / l;
* preoperative platelet content > 100 × 109 / l;
* preoperative hemoglobin> 120 g / l

Exclusion Criteria:

* pregnancy;
* planned valve surgery or surgery on the aorta;
* left main coronary artery stenosis> 75%;
* echocardiographic examination revealed moderate to severe mitral, tricuspid, or aortic regurgitation or stenosis;
* unstable or ongoing angina;
* recent (< 1 month) or ongoing acute myocardial infarction;
* use of sulfonylurea, theophylline or allopurinol;
* previous unusual response to an anesthetic agent;
* inclusion in other randomised controlled studies in the previous 30 days; (10)any general anesthesia performed in the previous 30 days;
* emergency operation (not scheduled);
* kidney or liver transplant in medical history, liver cirrhosis (Child B or C);
* chronic respiratory disease (such as chronic obstructive pulmonary emphysema)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
microRNA | 1h after isoflurane treatment(specimens of internal mammary artery and ascending aorta stump are saved)
NOS3 mRNA,mRNA levels of adhesion molecule selectin -E,vascular cell adhesion molecule -1,vascular endothelial growth factor -1,intercellular adhesion molecule,RhoA and ROK | 1h after isoflurane treatment(specimens of internal mammary artery and ascending aorta stump are saved)
phosphatidylinositol-3-kinase,alanine aminotransferase,endothelial nitric oxide synthase | 1h after isoflurane treatment(specimens of internal mammary artery and ascending aorta stump are saved)

SECONDARY OUTCOMES:
Change from microRNA | befor isoflurane treatment,1h,3h,5h after isoflurane treatment(central venous blood samples are drawn)
Change from ON content in serum,vascular cell adhesion molecule-1,intercellular adhesion molecules-1,adhesion molecule selectin-E,monocyte chemoattractant protein-1 and vascular endothelial growth factor-1 | befor isoflurane treatment,1h,3h,5h after isoflurane treatment(central venous blood samples are drawn)
Change from tumor necrosis factor-a,interleukin 1β,IL-6,IL-8 and IL-10 | befor isoflurane treatment,1h,3h,5h after isoflurane treatment(central venous blood samples are drawn)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang L, Wang CB, Li B, Lin DM, Ma J. RhoA/rho-kinase, nitric oxide and inflammatory response in LIMA during OPCABG with isoflurane preconditioning. J Cardiothorac Surg. 2019 Jan 25;14(1):22. doi: 10.1186/s13019-019-0835-9. PMID 30683137